CLINICAL TRIAL: NCT06914154
Title: Emulation of the SUMMIT Heart Failure Trial in Healthcare Claims Data
Acronym: DUP-SUMMIT
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-SUMMIT
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure With Preserved Ejection Fraction (HFPEF)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tirzepatide: Exposure group
  Interventions: Drug: Tirzepatide
- Placebo: Reference group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — New use of tirzepatide dispensing claim is used as the exposure.
  Groups: Tirzepatide
Drug: Placebo — New use of sitagliptin dispensing claim is used as the reference (active-comparator proxy for placebo).
  Groups: Placebo

SUMMARY:
Investigators are building an empirical evidence base for real-world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the SUMMIT trial described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. In addition to closely emulating the trial population, this study also evaluates outcomes in a broader, less restrictive cohort to enhance generalizability to patients typically encountered in routine clinical practice. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides guidance on the reference standard treatment effect estimate. However, failure to replicate RCT findings is not necessarily indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons, as the end points examined in the database study were partly only of exploratory nature in the trial. Moreover, divergence from these end points do not provide information on the validity of the original RCT finding.

The SUMMIT trial is a superiority trial that included an evaluation of the effect of tirzepatide, a dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (GLP-1) receptor agonist (RA), vs placebo on all-cause mortality or worsening heart failure events among individuals with heart failure with preserved ejection fraction.

The database study designed to emulate the type 2 diabetes mellitus (T2DM) subgroup of the SUMMIT trial will be a new-user active-comparative study, conducted using 2 national United States claims databases, where we compare the effect of tirzepatide vs sitagliptin, a dipeptidyl peptidase-4 inhibitor (DPP4i) on the composite end point of all-cause mortality or heart failure hospitalization. While the SUMMIT trial was conducted in participants with and without T2DM, both subgroups showed similar effect estimates in their results. Furthermore, while the trial compared tirzepatide vs placebo, we chose to use sitagliptin as an active-comparator proxy for placebo in the T2DM subgroup. Sitagliptin was specifically chosen because a major randomized controlled trial on cardiovascular outcomes demonstrated that the drug does not affect the cardiovascular outcomes under investigation. Furthermore, clinical guidelines during the study period recommended both drug classes under investigation as second- or third-line options for glucose lowering and were similarly costly.

ELIGIBILITY:
Eligible cohort entry dates:

Optum: Study period between May 13, 2022 to November 30, 2024 Marketscan: Study period between May 13, 2022 to December 31, 2023

FOLLOWING ELIGIBILITY OF THE SUMMIT TRIAL

Inclusion Criteria:

* ≥ 40 years old, male or female sex
* Chronic heart failure (NYHA Class II-IV) diagnosed for at least 3 months before Visit 1
* LVEF ≥50% demonstrated by echocardiogram performed at Visit 1 or within 6 months of Visit 1
* Structural heart disease
* Either one of: (1) eGFR <70 mL/min/1.73m2 at Visit 1, (2) HF decompensation within 12 months of Visit 1, defined as hospitalization for HF requiring IV diuretic treatment or urgent HF visit requiring IV diuretic treatment
* Stable dose of all concomitant HF medications (that is, beta blockers, ACEis, ARBs, and MRAs), except for oral diuretics, for at least 4 weeks prior to Visit 1 a
* If treated with oral diuretics, dose must be stable for at least 2 weeks prior to Visit 1 and throughout the screening period; volume control must be optimally achieved in the opinion of the investigator
* BMI ≥27.0 kg/m2 at Visit 1
* Type 2 diabetes mellitus trial subgroup

Exclusion Criteria:

* Myocardial infarction, coronary artery bypass graft surgery, or other major CV surgery/intervention, stroke or transient ischemic attack in past 90 days, or unstable angina pectoris in past 30 days, prior to Visit 1 or during screening
* Lung disease: pulmonary arterial hypertension, chronic thromboembolic pulmonary hypertension (CTEPH), or severe pulmonary disease including (COPD)
* Other medical conditions: severe anemia (hemoglobin level <9 g/dL) at Visit 1, untreated thyroid disease or TSH >4.0 mU/L at Visit 1, or significant musculoskeletal disease
* Orthopedic conditions that limit the ability to walk, such as severe arthritis in the leg, knee, hip injuries, hemiplegia, or amputation with artificial limb without stable prosthesis function
* Any condition that in the opinion of the investigator would interfere with the assessment of 6MWT
* LVEF <40% by local echocardiography documented any time within 2 years of Visit 1
* Acute decompensated HF (exacerbation of HF) requiring IV diuretics, IV inotropes, or IV vasodilators, or left ventricular assist device (LVAD) within 4 weeks prior to Visit 1, and/or during the screening period until randomization
* Impaired renal function, defined as eGFR <15 mL/min/1.73 m2 (CKD-EPI) or requiring dialysis at Visit 1
* Any one of the following: (1) Systolic blood pressure (SBP) ≥180 mmHg at Visit 1 (2) SBP >160 mmHg both at Visit 1 and at Visit 2 (3) Have symptomatic hypotension or SBP <100 mmHg at Visit 1 or Visit 2
* Atrial fibrillation or atrial flutter with a resting heart rate >110 bpm documented by ECG at Visit 1
* Cardiac amyloidosis or cardiomyopathy based on accumulation disease (for example, haemochromatosis, Fabry disease), muscular dystrophy, cardiomyopathy with reversible causes (for example, stress cardiomyopathy), hypertrophic obstructive cardiomyopathy or known pericardial constriction, or any severe (obstructive or regurgitant) valvular heart disease likely to lead to surgery during the study period
* Completed prior surgical treatment for obesity or had liposuction or abdominoplasty within 1 year prior to Visit 1. Participants who plan to have surgical treatment for obesity or liposuction or abdominoplasty during the duration of the study are excluded.
* Have type 1 diabetes mellitus
* For type 2 diabetes mellitus (1) Have uncontrolled diabetes requiring immediate therapy (such as diabetic ketoacidosis) at Visit 1 or Visit 2, in the judgement of the physician (2) Have had 1 or more events of severe hypoglycemia and/or 1 or more events of hypoglycemia unawareness within 6 months prior to Visit 1 (see Section 10.5.1.1 for definition of hypoglycemia) (3) Have a history of proliferative diabetic retinopathy, diabetic maculopathy, or severe nonproliferative diabetic retinopathy that requires acute treatment. Patients with T2DM should have had a dilated fundoscopic examination, performed by an ophthalmologist or optometrist, within 12 months of Visit 1 or prior to randomization (4) Treated with premix or prandial insulins or intensified insulin regimens (multiple daily injection with basal and prandial insulins or insulin pump therapy) at Visit 1
* History of acute or chronic pancreatitis or at high risk for acute pancreatitis (for example, serum triglyceride level >500 mg/dL
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease, or any of the following, as determined by the central laboratory during Visit 1: ALT or AST levels >2.5X the ULN for the reference range.
* Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome type 2
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous-cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) for less than 5 years
* Have a history of any other condition (such as known drug or alcohol abuse, diagnosed eating disorder, or other psychiatric disorder) that, in the opinion of the investigator, may preclude the participant from following and completing the protocol
* Have a known clinically significant gastric emptying abnormality (for example, severe diabetic gastroparesis or gastric outlet obstruction) or chronically take drugs that directly affect GI motility
* Treatment with any incretin, GLP-1 RA, or pramlintide in the 3 months prior to Visit 1
* Implantable cardioverter defibrillator (ICD) implantation within 1 month prior to Visit 1 or planned implantation during the course of the study
* Currently implanted left ventricular assist device (LVAD)
* Cardiac resynchronization therapy (CRT) implanted within 6 months prior to Visit 1 or planned implantation during the course of the trial
* Current use of medication associated with weight gain or weight loss, except when on stable dose for at least 3 months prior to Visit 1, and expected to be stable during the study period
* Pregnancy

RELAXING ELIGIBILITY OF THE SUMMIT TRIAL

Inclusion Criteria:

* Men or women ≥ 40 years old
* History of type 2 diabetes mellitus
* BMI ≥ 27.0 kg/m2
* Heart failure
* Preserved ejection fraction

Exclusion Criteria:

* Prior treatment with any GLP-1-RA
* History of type 1 diabetes mellitus
* End-stage renal disease or chronic or intermittent hemodialysis or peritoneal dialysis
* History of bariatric surgery
* History of nursing home admission
* Pregnant female or breast-feeding
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy
* Treatment with continuous subcutaneous insulin infusion
* Multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous-cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) for less than 5 years
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included individuals aged 40 years or older with heart failure with preserved ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 11265 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality or heart failure hospitalisation. | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs placebo (sitagliptin) on all-cause mortality or heart failure hospitalization in patients with heart failure with preserved ejection fraction when following the eligibility criteria of the SUMMIT trial.
Composite of all-cause mortality or heart failure hospitalization. | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs placebo (sitagliptin) on all-cause mortality or heart failure hospitalization in patients with heart failure with preserved ejection fraction when relaxing the eligibility criteria of the SUMMIT trial.

SECONDARY OUTCOMES:
Composite of all-cause mortality or all-cause mortality or a worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting). | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on composite of all-cause mortality or all-cause mortality or a worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting). in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting). | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting). in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Intravenous diuretic therapy in an urgent care setting | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on intravenous diuretic therapy in an urgent care setting in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Hospitalization for heart failure | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on hospitalization for heart failure in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
All-cause mortality | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on all-cause mortality in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Urinary tract infection | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on Urinary tract infection in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Serious bacterial infection | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on serious bacterial infection in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Gastrointestinal adverse effects | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on gastrointestinal adverse effects in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.

OTHER OUTCOMES:
Hernia | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on a negative control outcome of hernia in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.
Lumbar radiculopathy | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs placebo (sitagliptin) on a negative control outcome of lumbar radiculopathy in two populations: (1) patients meeting the eligibility criteria of the SUMMIT trial, and (2) a broader patient population when relaxing the eligibility criteria of the SUMMIT trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kruger N, Schneeweiss S, Fuse K, Matseyko S, Sreedhara SK, Hahn G, Schunkert H, Wang SV. Semaglutide and Tirzepatide in Patients With Heart Failure With Preserved Ejection Fraction. JAMA. 2025 Oct 14;334(14):1255-1266. doi: 10.1001/jama.2025.14092. PMID 40886075

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT06914154/Prot_SAP_001.pdf